CLINICAL TRIAL: NCT06607263
Title: Clinical Study to Evaluate the Efficacy of Rinsing With an Alcohol Free Mouthwash Containing CPC+Zn as Compared to Dental Flossing and to Rising With an Essential Oils Containing Alcohol Mouthwash in Reducing Dental Plaque and Gingivitis.
Brief Title: Comparative Study of CPC+Zn Mouthwash, Dental Floss, and Essential Oils Mouthwash on Plaque and Gingivitis Reduction
Acronym: PGMWI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2024-08-PG-MWI-BZ-CB
Record Dates: First submitted 2024-09-12; First posted 2024-09-23 (Actual); Last update posted 2025-04-14 (Actual); Status verified 2025-04

CONDITIONS: Gingival Bleeding; Plaque Induced Gingival Disease; Gingivitis and Periodontal Diseases
Keywords: dental plaque; gingivitis
MeSH Terms: conditions — Gingival Hemorrhage; Gingivitis; Periodontal Diseases; Dental Plaque | interventions — Dental Devices, Home Care; Toothpastes

STUDY DESIGN:
Intervention Model Description: This is a Phase III, randomized, controlled, double-blind, parallel-group clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this clinical trial, masking involves several key roles to ensure unbiased results. The Participant, Care Provider, Investigator, and Outcomes Assessor are all masked in this double-blind study. This means that the participants do not know which group they have been assigned to, the care providers administering the treatments are unaware of the specific products being used by each participant, the investigators conducting the study do not know the group assignments, and the outcomes assessors evaluating the results are blind to the treatment allocations. This comprehensive masking approach is designed to minimize any potential biases and maintain the integrity of the study results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPC + Zn mouthwash + Brushing (Experimental): A regimen composing a CPC + Zn mouthwash + Brushing with a fluoride toothpaste and a commercially available toothbrush
  Interventions: Drug: Mouthwash CPC+Zn+F; Drug: Toothpaste; Device: Toothbrush
- Essential oils mouthwash + Brushing (Active Comparator): A regimen composing a essential oils mouthwash + Brushing with a fluoride toothpaste and a commercially available toothbrush
  Interventions: Drug: Essential oils mouthrinse; Drug: Toothpaste; Device: Toothbrush
- Flossing + Brushing (Active Comparator): A regimen composing flossing + Brushing with a fluoride toothpaste and a commercially available toothbrush
  Interventions: Device: Dental floss; Drug: Toothpaste; Device: Toothbrush

INTERVENTIONS:
Drug: Mouthwash CPC+Zn+F — A mouthwash containing CPC + Zn and fluoride
  Other Names: CPC+Zn
  Arms: CPC + Zn mouthwash + Brushing
Drug: Essential oils mouthrinse — Essential oils mouthrinse
  Arms: Essential oils mouthwash + Brushing
Device: Dental floss — Dental floss
  Arms: Flossing + Brushing
Drug: Toothpaste — A commercially available fluoride toothpaste
Device: Toothbrush — A commercially available adult toothbrush

SUMMARY:
Clinical study evaluating the effectiveness of an alcohol-free mouthwash containing CPC+Zn compared to dental flossing and an essential oils-containing alcohol mouthwash in reducing dental plaque and gingivitis. This is a Phase III, single-center, double-blind trial with a parallel design. It involves 120 participants aged between 18 and 65, randomized into different groups, and spans 12 weeks.

DETAILED DESCRIPTION:
This clinical study aims to evaluate the efficacy of an alcohol-free mouthwash containing CPC (Cetylpyridinium Chloride) and Zinc (Zn) in reducing dental plaque and gingivitis compared to dental flossing and a mouthwash with essential oils in an alcohol base. It is a Phase III, randomized, double-blind, parallel-group trial involving 120 participants aged 18 to 65. Subjects will be divided into three groups-one using the CPC+Zn mouthwash, another using the essential oils mouthwash, and a control group using dental floss. Each group will also use a fluoride toothpaste and a soft-bristle toothbrush twice daily over 12 weeks. The primary efficacy variable is the reduction of gingival inflammation also Probing Depth, Bleeding on Probing, and a Plaque Index will be accessed. Subjects will undergo baseline, 4-week, and 12-week evaluations, with data analyzed using ANCOVA to assess the efficacy and safety of the products. Adverse events and compliance will be closely monitored, with strict confidentiality maintained for all participants. The study rigorous design aims to provide comprehensive insights into the effectiveness of these oral hygiene regimens.

ELIGIBILITY:
Inclusion Criteria:

* Availability for the duration of the study;
* Good general health (absence of any condition that, in the opinion of the Principal Investigator, might constitute a risk to the subject while participating in the study. Examples include heart problems, valve/hip replacements, etc);
* Willingness to provide information related to their medical history;
* ≥20 teeth with scorable facial and lingual surfaces; evidence of gingivitis;
* ≥10 bleeding sites based on the BI
* Initial mean gingivitis index of at least 1.5 as determined by the use of the Modified Gingival Index (MGI).
* Subjects without allergies to the products that are being tested;
* Informed Consent Form signed.

Exclusion Criteria:

* That received dental prophylaxis within 1 month prior to the Baseline visit;
* Need for antibiotics prior to dental treatment; use of antibiotics, anti-inflammatory or anticoagulant therapy during the three months prior to entry into the study;
* Usage of oral care products containing chemotherapeutic products within 2 weeks prior to Baseline;
* Use of smokeless tobacco;
* Any other condition that would make the volunteer inappropriate for the study.
* Oral pathology, chronic disease, or a history of allergy to testing products;
* Subject using anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory medication or daily analgesics within one month prior to the start of the study or scheduled to start such intake during the course of the study;
* Subject participating in any other clinical study;
* Subject pregnant or breastfeeding;
* Subject allergic to oral care products, personal care consumer products, or their ingredients;
* Ongoing use of medications known to affect the gingival tissues (i.e. calcium channel blockers, phenytoin, cyclosporine);
* Periodontal treatment 12 months before the beginning of the study;
* Current smokers and subjects with a history of alcohol or drug abuse;
* Subjects with orthodontic appliances or presence of fixed or removable prosthodontics dentures that may interfere with the evaluations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Modified Gingival Index | 12 weeks
  The Modified Gingival Index (MGI) is a clinical assessment tool used to evaluate the severity of gingivitis by measuring the extent of gingival inflammation. It categorizes gingival health on a scale from 0 to 4, where 0 signifies normal gingiva with no inflammation, and 4 indicates severe inflammation characterized by erythema, edema, and spontaneous bleeding.

SECONDARY OUTCOMES:
Turesky modification of Quigley-Hein Plaque Index | 12 weeks
  The Turesky modification of the Quigley-Hein Plaque Index is a method for assessing dental plaque accumulation by scoring plaque presence on six surfaces of each tooth on a scale from 0 to 5.
Bleeding on probing | 12 weeks
  Bleeding on probing (BOP) is a diagnostic technique used to assess gingival inflammation by gently probing the gum tissue; the presence of bleeding indicates inflammation and potential periodontal disease.
Probing depth | 12 weeks
  Probing depth measures the distance between the gingival margin and the bottom of the periodontal pocket using a calibrated periodontal probe, indicating the severity of periodontal disease.

CONTACTS AND LOCATIONS:
Overall Officials: Cassiano K Rosing, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No